CLINICAL TRIAL: NCT00828100
Title: Comparison of fluID Rapid Influenza and BinaxNOW® Influenza A & B
Brief Title: Comparison of Fluid Rapid Influenza and BinaxNOW Influenza A & B
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: Study currently suspended due to a lack of available funding.
Sponsor: Nanogen, Inc. (Industry)
Responsible Party: Philip Estes / Associate Director, Clinical, Nanogen, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FLU-13
Record Dates: First submitted 2009-01-20; First posted 2009-01-23 (Estimated); Last update posted 2009-03-06 (Estimated); Status verified 2009-03

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: fluID Rapid Influenza Test — The fluID™ Rapid Influenza Test is an in vitro diagnostic assay designed to be used with a reader for the qualitative detection of influenza type A and type B nucleoprotein antigens, and the differentiation of influenza type A subtypes A/H1 and A/H3 antigens associated with the seasonal influenza H1N1 and H3N2, in nasal swabs, nasopharyngeal swabs and nasal wash/aspirate specimens. The test is intended as an aid in the rapid, qualitative diagnosis of influenza type A and type B viral infections in patients symptomatic with influenza-like illness. The fluID™ Rapid Influenza Test is intended for use by a healthcare professional in a laboratory or Point-of-Care (POC) setting.
Device: BinaxNOW® Influenza A & B — The BinaxNOW Influenza A & B Test is an in vitro immunochromatographic assay for the qualitative detection of influenza A and B nucleoprotein antigens in nasopharyngeal (NP) swab and nasal wash/aspirate specimens. It is intended to aid in the rapid differential diagnosis of influenza A and B viral infections. Negative test results should be confirmed by culture.

SUMMARY:
The primary objective of this study is to compare the performance of the investigational fluid Rapid Influenza Test and the BinaxNOW® Influenza A & B Test in detecting influenza type A and influenza type B.

DETAILED DESCRIPTION:
The primary objective of this study is to compare the performance of the investigational fluID Rapid Influenza Test and the BinaxNOW® Influenza A & B Test in detecting influenza type A and influenza type B, with respect to fresh nasal wash / aspirate specimens collected from patients presenting with signs and symptoms of influenza-like illness (ILI). Specimens to be evaluated in this study will be enrolled in a concurrent clinical study per protocol FLU-05, entitled "Prospective Evaluation of the fluID Rapid Influenza Test". All subjects enrolled in the FLU-05 study will have consented to having their samples used in future investigations involving the fluID Test.

This study will be conducted during the 2008-2009 influenza season in North America and Hong Kong, which is anticipated to run from November 2008 to May 2009. Should the influenza season conclude in North America and Hong Kong prior to the attainment of the minimum target enrollment specified in the FLU-05 study, study sites in Australia will also be enlisted in order to enroll subjects; in such a case, enrollment will continue during the 2009 influenza season in these countries, which is anticipated to run from May through October, 2009.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects of any age;
2. Subjects presenting to the investigative site within 4 days of symptom onset, with:

   * Fever ≥ 38.0°C (100.4°F) if taken orally, or ≥ 38.5°C (101.2°F) if taken rectally; or a self-reported history of fever or feeling feverish (includes fever controlled by medication) in the absence of documented fever;
   * One or more respiratory symptoms of influenza-like illness which may include the following:
   * Sore throat
   * Runny or stuffy nose
   * Cough
   * One or more constitutional symptoms of influenza-like illness which may include the following:
   * Myalgia (aches and pains)
   * Headache
   * Fatigue
3. Subjects (or parent/guardian) willing and able to provide informed consent;
4. Subjects must be enrolled in Arm 3 of the FLU-05 clinical study.

Written subject informed consent for this study protocol must be obtained prior to study enrollment. Each subject (or parent or guardian) must personally sign and date the Subject Informed Consent Form prior to his/her participation in this clinical study.

Exclusion Criteria:

1. Subjects not presenting with at least three symptoms of influenza-like illness as outlined above.
2. Subjects who have received influenza antiviral medication or an investigational influenza drug treatment within the previous 30 days of study enrollment.
3. Subjects (children and adults) for whom the obtaining of aspirate samples is contraindicated or not possible.
4. Subjects with a medical condition that prevents nasal washes or aspirate samples from being obtained.
5. Active duty military personnel (participating military study sites only).
6. Subjects (or parent/guardian) unwilling or unable to provide informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 650 (Estimated)
Dates: Start 2009-02; Primary Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
Positive percent agreement and negative percent agreement for both influenza A and influenza B. | End of study

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Louisiana State University Health Sciences Center, Shreveport, Louisiana
  - Medical College of Wisconsin, Milwaukee, Wisconsin